CLINICAL TRIAL: NCT05401292
Title: Skin Preparation for Elective Foot and Ankle Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Kyle Schweser MD, Orthopaedic Trauma Surgeon, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2074962
Record Dates: First submitted 2022-02-23; First posted 2022-06-02 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Microbial Colonization; Foot and Ankle Disorders
MeSH Terms: conditions — Communicable Diseases | interventions — chlorhexidine gluconate; 2-Propanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iodine or Chlorhexidine Preparation (Active Comparator): Standard of care with only skin preparation of iodine or chlorhexidine solution prior to sterile draping before surgery.
  Interventions: Drug: Hibiclens
- Iodine or Chlorhexidine Scrub Brush Pre-Scrub with Isopropyl Alcohol and Chlorhexidine Soap (Active Comparator): In addition to standard of care skin preparation with iodine or chlorhexidine solution prior to sterile draping, patients will also receive an additional "pre-scrub" with isopropyl alcohol and chlorhexidine soap. The operative extremity will be scrubbed for 2 minutes with chlorhexidine soap with a scrub brush until the entire extremity is covered. Isopropyl alcohol will then be wiped onto the skin with a gauze and allowed to evaporate (dry).
  Interventions: Drug: Hibiclens; Drug: Isopropyl Alcohol 70% Topical Application Solution

INTERVENTIONS:
Drug: Hibiclens — antiseptic/antimicrobial skin cleanser for skin wound and general skin cleansing
Drug: Isopropyl Alcohol 70% Topical Application Solution — First aid antiseptic
  Arms: Iodine or Chlorhexidine Scrub Brush Pre-Scrub with Isopropyl Alcohol and Chlorhexidine Soap

SUMMARY:
Surgical site infections (SSIs) make about 31% of all nosocomial infections and they are the most common hospital-acquired infection. For foot and ankle elective interventions, SSI rate is reported between 0.4% and 3.6%. This study will investigate the effectiveness of skin cleaning with isopropyl alcohol and scrubbing with chlorhexidine soap before standard skin preparation in reducing microbial load and surgical site infections for elective foot and ankle surgeries. Current standard of care includes skin preparation with iodine or chlorhexidine solution prior to sterile draping and the start of surgery. Standard of care will be applied to all patients. The use of an additional "pre-scrub" with isopropyl alcohol and scrubbing with chlorhexidine soap will be applied to the experimental group. The control group will receive only the standard of care skin preparation with iodine or chlorhexidine solution prior to draping.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective foot and ankle surgeries
* age over 18

Exclusion Criteria:

* trauma as the indication for surgery
* open injuries
* non-elective procedures
* amputations
* prior surgical site infection through the planned incision
* pregnancy. All potential participants of child-bearing potential follow the standard pre-operative protocol to ensure they are not in pregnant status prior to SOC surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 90 days
  rate of surgical site infection (SSI) and wound complications following skin preparation for surgery. Measured by the number of surgical site infections in the total population of patients in the cohort

SECONDARY OUTCOMES:
Microbial Load | 90 days
  effectiveness of reducing microbial load. Comparing original microbial load to final microbial load (CFU/g)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided